CLINICAL TRIAL: NCT07369622
Title: A Prospective Interventional Study Comparing Genotype-Guided Therapy Versus Usual Care to Prevent Severe Cutaneous Adverse Reactions Associated With Allopurinol and Carbamazepine in Vietnam
Brief Title: HLA-B*58:01-Guided Therapy for Gout: Effectiveness, Safety, and Cost-Effectiveness
Acronym: HLA-SCREEN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLA-GOUT-SCARS-2026; HPMU-HLA-GOUT (Other: Hai Phong University of Medicine and Pharmacy (HPMU))
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Gout Initiating Urate-loweringUrate-lowering Therapy; Gout Arthritis; Gout and Hyperuricemia
Keywords: HLA-B*58:01; HLA genotyping; Pharmacogenomics; Allopurinol; febuxostat; Pharmacogenetic screening; Severe cutaneous adverse reactions (SCARs); Stevens-Johnson syndrome (SJS); Toxic epidermal necrolysis (TEN); Cost-effectiveness analysis
MeSH Terms: conditions — Arthritis, Gouty; Gout; Hyperuricemia; Stevens-Johnson Syndrome | interventions — Allopurinol; Febuxostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HLA-B*58:01 Negative: Allopurinol (Active Comparator): Participants test negative for HLA-B*58:01 and initiate allopurinol as first-line urate-lowering therapy. Follow-up for 12 months with visits at baseline, 1, 3, 6, and 12 months to assess serum urate control, gout flares, and safety (including active surveillance for SCARs and routine liver/kidney function monitoring).
  Interventions: Diagnostic Test: HLA-B*58:01 Genotyping; Drug: Allopurinol Tablet
- HLA-B*58:01 Positive: Febuxostat (Active Comparator): Participants test positive for HLA-B*58:01 and receive febuxostat as an alternative urate-lowering therapy to avoid allopurinol-associated SCAR risk. Follow-up for 12 months with visits at baseline, 1, 3, 6, and 12 months to evaluate serum urate response, gout flares, and safety outcomes.
  Interventions: Diagnostic Test: HLA-B*58:01 Genotyping; Drug: Febuxostat
- No HLA-B*58:01 Testing: Febuxostat (Active Comparator): Participants do not undergo HLA-B*58:01 testing and are treated directly with febuxostat as urate-lowering therapy under routine clinical practice. Follow-up for 12 months with visits at baseline, 1, 3, 6, and 12 months to assess effectiveness (serum urate control, gout flares) and safety (including SCAR surveillance and laboratory monitoring).
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Diagnostic Test: HLA-B*58:01 Genotyping — Whole-blood sample is collected for HLA-B58:01 genotyping using a PCR-based assay with allele-specific primers. Results are classified as HLA-B58:01 positive or negative and are used to guide urate-lowering therapy selection (allopurinol for negative; febuxostat for positive).
  Other Names: HLA-B*5801 test; PCR-based HLA-B*58:01 typing
  Arms: HLA-B*58:01 Negative: Allopurinol; HLA-B*58:01 Positive: Febuxostat
Drug: Allopurinol Tablet — Oral allopurinol is initiated as urate-lowering therapy in participants who are HLA-B*58:01 negative. Dosing and titration follow routine clinical practice with consideration of kidney function and serum urate targets. Participants are followed for 12 months with scheduled visits to assess serum urate control, gout flares, and safety outcomes including active surveillance for severe cutaneous adverse reactions (SCARs).
  Other Names: Xanthine oxidase inhibitor
  Arms: HLA-B*58:01 Negative: Allopurinol
Drug: Febuxostat — Oral febuxostat is used as an alternative urate-lowering therapy for participants who are HLA-B*58:01 positive to avoid allopurinol-associated SCAR risk, and for a comparison cohort treated without HLA testing. Participants are followed for 12 months with scheduled visits to evaluate serum urate response, gout flares, and safety (including SCAR surveillance and routine liver/kidney function monitoring).
  Other Names: Xanthine oxidase inhibitor
  Arms: HLA-B*58:01 Positive: Febuxostat; No HLA-B*58:01 Testing: Febuxostat

SUMMARY:
Severe cutaneous adverse reactions (SCARs), such as Stevens-Johnson syndrome/toxic epidermal necrolysis (SJS/TEN) and drug reaction with eosinophilia and systemic symptoms (DRESS), are rare but life-threatening complications that can occur after starting allopurinol for gout. The HLA-B58:01 allele is a strong genetic risk factor for allopurinol-associated SCARs in Asian populations. This study evaluates the feasibility and clinical value of HLA-B58:01 screening before first-time allopurinol use in Vietnamese adults with gout.

Adults (≥18 years) diagnosed with gout (ACR/EULAR 2020 criteria) and initiating urate-lowering therapy will be enrolled at Hai Phong International General Hospital (January 2025-June 2027). Participants who undergo HLA-B58:01 genotyping (PCR-based assay) will be treated according to test results: HLA-B58:01 negative participants receive allopurinol; HLA-B58:01 positive participants receive febuxostat. A comparison group consists of patients treated with febuxostat without HLA testing. Participants will be followed for 12 months with assessments at baseline, 1, 3, 6, and 12 months to monitor serum uric acid, gout flares, and safety outcomes (SCARs and other adverse events, including liver and kidney function). The study also includes an economic evaluation to estimate the cost-effectiveness of HLA-B58:01 screening for preventing SCARs and optimizing gout treatment.

DETAILED DESCRIPTION:
Background and rationale: Allopurinol is a first-line urate-lowering therapy for gout but is a leading cause of severe cutaneous adverse reactions (SCARs), including SJS/TEN and DRESS. These reactions carry substantial morbidity, mortality, and healthcare costs. Genetic susceptibility-particularly carriage of HLA-B*58:01-has been consistently associated with allopurinol-induced SCARs, and pre-treatment HLA screening has reduced SCARs in several Asian settings. However, implementation evidence in Vietnam remains limited. This study is designed to generate local clinical and economic evidence to support an HLA-guided prescribing strategy.

Study objectives:

Describe the prevalence of HLA-B*58:01 among adult Vietnamese patients with gout initiating allopurinol for the first time.

Compare effectiveness and safety outcomes between an HLA-guided strategy (allopurinol for HLA-B58:01 negative; febuxostat for HLA-B58:01 positive) and a non-tested febuxostat strategy.

Evaluate the cost-effectiveness of HLA-B*58:01 screening in preventing SCARs and informing treatment selection.

Study setting and timeframe: Single-center study at Hai Phong International General Hospital, Vietnam, from January 2025 to June 2027.

Design overview:

Descriptive cross-sectional component to estimate HLA-B*58:01 positivity among tested, eligible patients.

Prospective comparative follow-up over 12 months to evaluate real-world effectiveness and safety of urate-lowering strategies.

Cost-effectiveness analysis using direct medical costs.

Participants:

Inclusion criteria include age ≥18 years, gout diagnosis according to ACR/EULAR 2020, first-time indication for allopurinol, and willingness to provide clinical data and undergo HLA testing (for tested groups). Exclusion criteria include prior allopurinol exposure or prior allopurinol hypersensitivity, severe comorbid/complex conditions likely to confound treatment (e.g., end-stage kidney disease, advanced malignancy, bone marrow transplantation, current immunosuppression), or inability to adhere to follow-up.

Interventions/Groups:

Group 1 (HLA-B*58:01 negative; allopurinol): participants tested negative and start allopurinol.

Group 2 (HLA-B*58:01 positive; febuxostat): participants tested positive and use febuxostat as an alternative.

Group 3 (No HLA test; febuxostat): participants treated directly with febuxostat without HLA testing.

Procedures and follow-up schedule:

HLA-B*58:01 genotyping is performed on whole blood using PCR with sequence-specific primers; results are classified as positive or negative.

Follow-up visits at baseline, 1, 3, 6, and 12 months.

Clinical and laboratory monitoring includes serum uric acid and safety labs (AST/ALT, creatinine/eGFR) at predefined time points; gout flare frequency and severity are recorded (including pain assessment using VAS).

SCARs are actively surveilled and clinically diagnosed; supportive laboratory findings include eosinophilia and hepatic/renal involvement when applicable.

Outcome measures:

Genetic outcome: prevalence of HLA-B*58:01 positivity among tested participants.

Effectiveness outcomes: change in serum uric acid over time; proportion achieving target uric acid control; frequency and severity of gout flares during follow-up.

Safety outcomes: incidence of SCARs (SJS, TEN, DRESS); other adverse events including liver enzyme elevation and renal function deterioration; mild hypersensitivity manifestations (e.g., pruritus, urticaria).

Economic outcomes: direct costs of HLA testing, drug therapy, laboratory monitoring, and SCAR management (hospitalization, medications, procedures, investigations). Cost-effectiveness metrics include the cost per unit of SCAR risk reduction and comparative total costs between strategies.

Sample size considerations:

A descriptive sample size is calculated to estimate HLA-B*58:01 prevalence, and a comparative sample size is calculated for effectiveness/safety comparisons between allopurinol and febuxostat strategies; the planned comparative cohort is approximately 114 participants per treatment strategy group.

Ethics:

The study is conducted in accordance with the Declaration of Helsinki and Good Clinical Practice. Participants provide informed consent; confidentiality is maintained; participants may withdraw at any time without affecting standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.

Diagnosis of gout according to the 2020 ACR/EULAR classification criteria.

Indicated for initiation of urate-lowering therapy (ULT) and allopurinol-naïve (no prior allopurinol exposure).

Able and willing to comply with scheduled follow-up visits (baseline, Months 1, 3, 6, and 12).

Provides written informed consent for participation.

For the genotyping arms: provides consent for blood sampling and HLA-B*58:01 genotyping.

Exclusion Criteria:

* Prior use of allopurinol or history of hypersensitivity reaction to allopurinol.

Known hypersensitivity to febuxostat (for participants who would receive febuxostat).

Current or recent severe skin reaction (suspected/confirmed SCAR) from any cause.

End-stage kidney disease requiring dialysis or kidney transplantation.

Severe hepatic impairment or active severe liver disease (e.g., AST/ALT >3× ULN at baseline).

Severe uncontrolled medical conditions that, in the investigator's judgment, could interfere with treatment or follow-up (e.g., decompensated heart failure, active malignancy requiring intensive treatment).

Use of systemic immunosuppressive therapy (e.g., high-dose corticosteroids, biologics, chemotherapy) at enrollment.

Pregnancy or breastfeeding.

Participation in another interventional clinical study that could affect the outcomes of this study.

Inability to provide informed consent or inability to adhere to study procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Target Serum Uric Acid <5.0 mg/dL (≈300 µmol/L) | At Month 12 after initiation of urate-lowering therapy
  Serum uric acid is measured by venous blood sampling using an automated biochemistry analyzer at baseline and follow-up visits (1, 3, 6, and 12 months). The primary endpoint is the proportion of participants who achieve the target serum uric acid level <5.0 mg/dL (approximately <300 µmol/L) at the 12-month visit.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in the primary publication, including demographics, baseline clinical characteristics, HLA-B*58:01 status (positive/negative), treatment assignment, longitudinal serum urate values, gout flare outcomes, adverse events (including SCARs), and cost variables. No direct identifiers will be shared; no raw genetic sequence data will be provided.
  Supporting Information to be Shared
  Study protocol, statistical analysis plan, data dictionary, and analytic code.
  Time Frame
  Beginning 6 months after publication of the primary results and ending 5 years thereafter.
  Access Criteria
  Researchers who provide a methodologically sound proposal may request access. Proposals will be reviewed by the study team and approved in accordance with institutional policies and applicable regulations. Access will be granted after signing a data use agreement. Data will be shared for the purpose of scientific research only, and recipien
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of the primary results and ending 5 years thereafter.
Access Criteria: De-identified individual participant data (IPD) that underlie the results reported in the primary publication, along with the study protocol (and SAP/analytic code if selected), will be available upon reasonable request. Requests may be submitted by qualified researchers with a methodologically sound proposal to the corresponding author. Proposals will be reviewed by the study team and approved in accordance with institutional policies and applicable regulations. Access will be granted after execution of a data use agreement. Data will be provided in de-identified form; no direct identifiers will be shared and recipients must not attempt re-identification.